CLINICAL TRIAL: NCT05734183
Title: Effects of Immersive Multisensory Stimulation in Disorders of Consciousness
Brief Title: Multisensorial IMmersive Experiences (MIME) in Disorders of Consciousness
Acronym: MIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, PADUA LUCA, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0038186/21
Record Dates: First submitted 2023-02-06; First posted 2023-02-17 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Disorder of Consciousness; Acquired Brain Injury
Keywords: Disorder of Consciousness; Acquired Brain Injury; Sensory stimulation
MeSH Terms: conditions — Consciousness Disorders; Brain Injuries | interventions — MIME protocol; Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MIME Group (Experimental): Stimulation with MIME will be performed in a large ad hoc room in which video images will be projected on three walls. The patient will be positioned in the center of the room, 3 meters from the front wall, with the back of the bed tilted at a 45-degree angle, so as to obtain a truly immersive view covering the entire 220-degree field of view. Audio stimulation will be achieved through two speakers located at the sides of the room, with the low frequencies reinforced by a subwoofer. The average sound intensity recorded from the patient's position will be 81 db average (maximum 87, minimum 69).
  Patients will undergo treatment with MIME once a day for five consecutive days, for a total of two weeks (10 sessions), in addition to conventional treatment.
  Interventions: Other: MIME
- MIME + tDCS Group (Active Comparator): Simultaneously with MIME treatment, patients will undergo transcranial direct current stimulation (tDCS). Stimulation with tDCS will begin 5 minutes after the start of resting phase 1, and the electrodes will be placed as follows: the 5×4 anode (about 20 cm2) will be placed on the left dorsolateral prefrontal area; the reference electrode, 6x5 (about 30 cm2), will instead be placed on the upper arm, specifically at the level of the right deltoid muscle, contralateral to the active electrode. Current will be applied at an intensity of 2 mA, for 20 minutes a day for 2 weeks, five days a week, for a total of 10 sessions. The current density will be kept below the safe limits reported in the literature.
  Interventions: Other: MIME + tDCS

INTERVENTIONS:
Other: MIME — Multisensorial IMmersive Experiences
  Arms: MIME Group
Other: MIME + tDCS — Multisensorial IMmersive Experiences plus transcranial direct current stimulation
  Arms: MIME + tDCS Group

SUMMARY:
Disorder of consciousness (DoC) is a state in which consciousness is altered because of brain damage and can occur under a variety of conditions: in fact, the most frequent causes of DoC are vascular disease, head trauma, and cerebral hypoxia. DoCs result from the loss of regulation of neural function of the two components of consciousness, alertness and awareness. Depending on the patient's behavior and responsiveness, DoCs can be identified in different states, from coma to persistent vegetative state (VS) to intermittent minimally conscious state (MCS). Regarding the prognosis of recovery, in patients with DoC the chance of having functional improvement decreases with time, although some positive functional changes have been observed in chronic patients. Therapies for DoC include some drugs, such as dopaminergic, GABAergic and amantadine drugs, which work to facilitate the recovery of consciousness. Neurorehabilitation, however, seems to be the most recognized intervention that aims to strengthen, in uninjured brain regions, the spontaneous neuroplasticity that occurs to compensate for lost function.

Simultaneous stimulation of multiple senses, such as hearing, sight and smell, provides the neural network with more stimuli that are more effective than a single stimulus. In fact, multisensory stimuli can more easily activate attention because cortical processing is predominantly multimodal. As for content, it would seem that those with autobiographical and emotionally salient character could engage multiple brain networks and have priority access to attention. Numerous trials show that stimulus-containing content led to increased behavioural activity, improving self-awareness in patients with DoC.

Considering that a communication system that can combine both visual and auditory channels proves to be more effective than a "single-sense" channel, multisensory stimulation is likely to provide simultaneous activation of different brain areas by enhancing plasticity processes. Furthermore, the intensity of stimulation could be one of the main variables with greater impact on the patient: in fact, higher intensity would correspond to a greater effect on the brain.

DETAILED DESCRIPTION:
It can be hypothesized that sensory stimulation, or "Multisensorial IMmersive Experiences" (MIME), enhanced by high-quality video images, a larger screen size, and qualitatively better sound, may have a greater impact on the patient than the same image or video played on a small screen.

The purpose of the study is to evaluate (i) whether MIMEs can clinically modify the vigilance of DoC patients during administration; (ii) whether there is SNA activation during the administration of MIMEs; and (iii) whether patients treated daily with MIMEs have any benefits in terms of vigilance modification.

Twenty patients of both sexes with DoC will be recruited, evaluated and treated at the UOC of High Intensity Neurorehabilitation at the Fondazione Policlinico Universitario Gemelli IRCCS in Rome.

All study participants will undergo MIME treatment once a day for 5 days a week, for a total of 10 sessions. Patients will perform, in addition to MIME therapy, conventional rehabilitation as a daily routine. Patients will be divided into two groups: one part will perform MIME treatment concurrently with transcranial direct current stimulation (tDCS, G-Mt) and as many will undergo MIME treatment alone (G-M), as described below. In the case of epileptic subjects, these due to contraindications to tDCS may be subjected to MIME therapy only.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 90 years Patients who have been in a coma state and have alterations in consciousness Patients who are not responsive to rehabilitative treatment of disorders of consciousness, such as environmental stimulation, non-invasive brain stimulation, or drug treatment.

Clinical stability Ability of caregiver/legal guardian to understand and sign informed consent

Exclusion Criteria:

Taking medications that interfere with membrane conductivity (e.g., calcium channel blockers, antiepileptic drugs).

Psychiatric or other medical conditions Failure to sign informed consent The presence of a history of epilepsy and/or taking antiepileptic therapy is an exclusion criterion for assignment to the MIME+tDCS group.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Coma Recovery Scale-r (CRS-r) | Change from baseline CRS-r at 2 weeks
  CRS-r is an assessment tool that examines 6 functions: auditory, visual, oral-verbal motor, communicative, and vigilance.
  Its different items are organized hierarchically (low scores represent reflex activities, high scores describe cognitively mediated behaviors).
  For each function examined, the diagnosis of Vegetative State, Minimal Consciousness State, Emergence from Minimal Consciousness State can be made.

SECONDARY OUTCOMES:
Electrodermal Activity (EDA) | Change from baseline EDA at 2 weeks
  The E4 wearable medical device (Empatica, EDA) will be used to assess the electrodermal activity (EDA).
  Fluctuations in some electrical properties of the skin will be recorded; the online software Empatica (https://www.empatica.com/en-eu/) will then export the recorded data.
  A higher EDA value corresponds to a higher stress level.
Heart Rate Variability (HRV) | Change from baseline HRV at 2 weeks
  HRV, that is, the assessment of heart rate variability, is evaluated using an electrocardiographic (ECG) device with normal surface electrodes applied at the level of the heart and special software for data analysis.
Level of Cognitive Functioning (LCF) | Change from baseline LCF at 2 weeks
  LCF is a tool that assesses the level of cognitive and behavioural recovery. It consists of 7 items ranging from 1=no response to 8=final-appropriate.
Disability Rating Scale (DRS) | Change from baseline DRS at 2 weeks
  DRS is an assessment tool for level of consciousness and functional recovery. It consists of four domains:
  (i) Vigilance, awareness and responsiveness (0 to 12 points) (ii) Cognitive ability for self-care activities (0 to 9 points) (iii) Functional level (0 to 5 points) (iv) employability (0 to 3 points). A higher score corresponds to greater disability. The overall score ranges from 0 to 30 and allows the identification of 10 categories ranging from category 1 (no disability) to category 10 (death).
Cognitive Reserve Index questionnaire (CRIq) | Assess CRIq at baseline
  The CRIq questionnaire evaluates the cognitive reserve of an individual by means of the compilation of information relating to his or her entire adult life. The questionnaire is divided into 3 sections: CRI-Education, CRI-WorkingActivity, CRI-LeisureTime.
  CRI-Education: this section records the level of education reached by an individual during his/her life. For each school year successfully completed, 1 point is assigned, whereas 0.5 points are assigned for each year that the individual was forced to repeat.
  CRI-WorkingActivity: this section records the type and number of years of work carried out by an individual.
  CRI-LeisureTime: this section refers to all of those activities that are normally carried out before or after the person concerned goes to work or school. The items included indicate the activity for which it is necessary to estimate the frequency within the given time interval.
Lifetime Physical Activity Questionnaire (LTPAQ) | Assess LTAQ at baseline
  LTPAQ is a questionnaire that collects information pertaining lifetime PA. It consists of three different sections: (i) Occupational and Volunteer Activities, (ii) Family Activities, and (iii) Exercise and Sports Activities.
  (i) Occupational and Volunteer Activities, the individual must indicate those jobs, paid or voluntary, that he/she has held for at least 8 hours per week for 4 months of the year.
  (ii) Family Activities, each individual must indicate the household, do-it-yourself, and gardening activities performed over a lifetime, for at least 7 hours per week for 4 months per year. Childcare is included in this section and sedentary activities are excluded.
  (iii) Exercise & Sports Activities, each individual must list all physical activity or sports he/she has done throughout his/her life since childhood, reporting activities he/she has done at least 2 hours per week for 4 months per year.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Padua, MD, phD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No